CLINICAL TRIAL: NCT07258056
Title: GUidance In Prostate Cancer DEtection With 18F-PSMA-1007-PET/MRI and Targeted Biopsies (GUIDE PSMA PET/MRI)
Brief Title: GUidance In Prostate Cancer DEtection With 18F-PSMA-1007-PET/MRI and Targeted Biopsies
Acronym: GUIDE PSMA PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mads Ryo Jochumsen (Other)
Responsible Party: Sponsor-Investigator, Mads Ryo Jochumsen, MD, Ph.D., Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-109-25
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: PSMA; PET/MRI; Prostate cancer; biopsy guidance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA-guided and systematic biopsies (Experimental): Both PSMA-guided and systematic biopsies are performed
  Interventions: Diagnostic Test: PSMA-guided and systematic biopsies

INTERVENTIONS:
Diagnostic Test: PSMA-guided and systematic biopsies — Both PSMA-guided and systematic biopsies are performed

SUMMARY:
The goal of this clinical study is to test the performance of PSMA PET/MRI-guided biopsies against systematic biopsies in men with negative MRI scan (PI-RADS 1-2) of the prostate with continuous suspicion of clinically significant prostate cancer (csPCa) due to PSAd > 0.20. The main questions it aims to answer are:

Can biopsies safely be avoided at PRIMARY score 1-2 without missing csPCa? Does targeted PSMA PET/MRI-guided biopsies have a higher detection rate of csPCa compared to systematic biopsies?

Participants will undergo both transperineal MRI/ultrasound fusion target biopsies from PRIMARY score 3-5 lesions on PSMA PET and systematic biopsies irrespective of the PRIMARY-lesion.

ELIGIBILITY:
Inclusion Criteria:

* PSAdensity > 0.20
* Negative MRI (PI-RADS 1-2) or negative biopsy from MRI-target
* MRI within 6 months
* Read and understand danish
* Expected remaining lifetime > 10 years

Exclusion Criteria:

* Known prostate cancer
* MRI contraindications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of clinically significant prostate cancer (csPCa) for PSMA guided biopsies vs systematic biopsies | From enrollment to pathology report is ready, assessed up to 2 years
  CsPCa is defined as "International Society of Urological Pathology" (ISUP) grade ≥ 2.
  The ISUP grade scale ranges from 1 to 5, where grade 1 is low-risk / indolent / non-significant prostate cancer and grade 5 is the most aggressive prostate cancer form with worse outcome.

SECONDARY OUTCOMES:
High negative predictive value for having csPCa in case of PRIMARY 1-2 (and PI-RADS 1-2) | From enrollment to pathology report, assessed up to 2 years
  A high negative predictive value for having csPCa in case of PRIMARY 1-2 (and PI-RADS 1-2) means that biopsies can safely be avoided in patients with PRIMARY 1-2 lesions only.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N, Aarhus
  - Goedstrup Hospital, Herning, Herning

IPD SHARING:
Plan to Share IPD: No
Relevant data from the study will be made avilable and published, but the investigators do not have permission to share individual participant data with external researchers.